CLINICAL TRIAL: NCT02046603
Title: Open-Label, Phase IIIb Study to Evaluate the Efficacy and Safety of Subcutaneous (SC) Tocilizumab Monotherapy or Combination Therapy With Methotrexate (MTX) or Other Non-Biologic Disease Modifying Anti-Rheumatic Drugs (DMARDs) in Patients With Active Rheumatoid Arthritis (RA) Who Have an Inadequate Response to Current Non-Biologic DMARD Therapy or the First Anti-Tumour Necrosis Factor (Anti-TNF) Biologic Agent
Brief Title: A Study of Tocilizumab (RoActemra/Actemra) in Monotherapy or in Combination With Methotrexate or Other Non-Biologic DMARDs in Participants With Active Rheumatoid Arthritis and an Inadequate Response to Current Non-Biologic DMARD Therapy or the First Anti-TNF Biologic Agent
Acronym: ACT-MOVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28641; 2013-000054-22 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents; Adrenal Cortex Hormones; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab Monotherapy (Experimental): Participants will receive a weekly SC injection of tocilizumab 162 mg as monotherapy for 52 weeks.
  Interventions: Drug: Tocilizumab
- Tocilizumab in Combination With Methotrexate or Other DMARDs (Experimental): Participants will receive a weekly SC injection of tocilizumab 162 mg in combination with methotrexate or other non-biologic DMARDs for 52 weeks.
  Interventions: Drug: Tocilizumab; Drug: DMARDs; Drug: Oral Corticosteroids; Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 162 mg will be administered once a week by SC injection and as a single fixed dose, irrespective of body weight, for the treatment duration of 52 weeks.
  Other Names: RoActemra, Actemra
Drug: DMARDs — Treatment with non-biologic DMARDs, at a stable dose that was initiated at least 4 weeks prior to baseline, is permitted during the study. The study protocol does not specify any particular therapy.
  Arms: Tocilizumab in Combination With Methotrexate or Other DMARDs
Drug: Oral Corticosteroids — Stable oral corticosteroids doses (≤10 mg/day prednisone or equivalent) are allowed. The study protocol does not specify any additional detail on types of oral corticosteroids.
  Arms: Tocilizumab in Combination With Methotrexate or Other DMARDs
Drug: Methotrexate — Methotrexate per investigator's discretion.
  Arms: Tocilizumab in Combination With Methotrexate or Other DMARDs

SUMMARY:
This open-label study will evaluate the efficacy and safety of tocilizumab as monotherapy or in combination with methotrexate or other non-biologic disease modifying anti-rheumatic drugs (DMARDs) in participants with active rheumatoid arthritis (RA) and an inadequate response to current non-biologic DMARD therapy or the first anti-tumour necrosis factor (anti-TNF) agent. Participants will receive tocilizumab 162 milligrams (mg) subcutaneously once a week for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Active RA according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria
* Participants who have an inadequate response to current non-biologic DMARD therapy or the first anti-TNF agent (in monotherapy or in combination with MTX or other non-biologic DMARDs). Inadequate response to anti-TNF treatment is defined as DAS28 score improvement of less than 1.2 or participants achieving a DAS28 score improvement of 1.2 but not achieving low disease activity (current DAS28-ESR above 3.2) according to a treat-to-target strategy and have not been previously exposed to treatment with tocilizumab. Inadequate response to non-biologic DMARD therapy will be assessed according to local guidelines and the participants will need to be eligible for biologic therapy according to local guidelines
* Oral corticosteroids (≤10 mg/day prednisone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs; up to recommended dose) are permitted if on stable dose regimen for greater than or equal to [≥] 4 weeks prior to baseline
* Permitted non-biologic DMARDs are allowed if on stable dose for at least 4 weeks prior to baseline
* Receiving treatment on an outpatient basis, not including tocilizumab
* Females of childbearing potential and males with female partners of childbearing potential must agree to use reliable means of contraception as defined by protocol during the study and for at least 3 months following the last dose of tocilizumab

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline
* Rheumatic autoimmune disease other than RA
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16
* Prior history of or current inflammatory joint disease other than RA
* Exposure to tocilizumab either intravenous or SC at any time prior to baseline
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Known active current or history of recurrent infections
* Major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years
* Positive for hepatitis B or hepatitis C virus infection
* Primary or secondary immunodeficiency (history of or currently active)
* Pregnant or lactating women
* Inadequate hematologic, renal or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United Kingdom (38):
  - Aberdeen Royal Infirmary, Aberdeen
  - Christchurch Hospital; Rheumatology, Bournemouth
  - Royal Sussex County Hospital; Clinical Investigation Research Unit, Brighton
  - Queens Hospital, Burton-on-Trent
  - West Suffolk Hospital, Bury Saint Edmonds
  - Addenbrooke'S Hospital; Rheumatology Research Unit, Cambridge
  - Cannock Chase Hospital; Rheumatology, Cannock
  - University Hospital of Wales; Dept of Rhematology, Cardiff
  - Broomfield Hospital, Chelmsford
  - Countess of Chester Hospital; Dept of Rheumatology, Chester
  - Dewsbury & District Hospital; Dept of Rheumatology, Dewsbury
  - Russells Hall Hospital; Rheumatology Department, Dudley
  - Ninewells Hospital, Dundee
  - Eastbourne District General Hospital; Dept of Rheumatology, Eastbourne
  - Western General Hospital; Pharmacy Department, Edinburgh
  - Gartnavel General Hospital; Rheumatology, Glasgow
  - Diana Princess of Wales Hosp., Grimsby
  - Princess Alexandra Hospital, Harlow
  - Northwick Park Hospital, Harrow
  - Hemel Hempstead General Hospital; Rheumatology Dept, Hemel Hempstead
  - Hull Royal Infirmary; Rheumatology Department, Hull
  - Llandudno General Hospital, Llandudno
  - Whipps Cross Hospital; Rheumatology Dept, London
  - Royal Free Hospital; Department of Rheumatology, London
  - Maidstone Hospital; Dept of Rheumatology, Maidstone
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital; Dept of Rheumatology, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Norfolk & Norwich Hospital; Rheumatology, Norwich
  - Integrated Care Centre, Oldham
  - Solihull Hospital, Solihull
  - Haywood Hospital; Staffordshire Rheumatology Centre, Stoke-on-Trent
  - Great Western Hospital; Dept of Rheumatology, Swindon
  - Torbay Hospital; Dept of Rhematology, Torquay
  - Royal Cornwall Hospital; Rhuematololgy Dept, Truro
  - Warrington Hospital, Warrington
  - Wrightington Hospital; Rheumatology, Wigan
  - Wishaw General Hospital, Wishaw

REFERENCES:
- [Derived] Isaacs JD, Salih A, Sheeran T, Patel YI, Douglas K, McKay ND, Naisbett-Groet B, Choy E. Efficacy and safety of subcutaneous tocilizumab in rheumatoid arthritis over 1 year: a UK real-world, open-label study. Rheumatol Adv Pract. 2019 Apr 19;3(1):rkz010. doi: 10.1093/rap/rkz010. eCollection 2019. PMID 31431998
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 participants were enrolled. One participant who did not receive a dose of tocilizumab was excluded from the full analysis set (FAS) and the results are reported for 161 participants.
Groups:
- Tocilizumab Monotherapy: Participants received a weekly subcutaneous (SC) injection of tocilizumab 162 milligrams (mg) as monotherapy for 52 weeks.
- Tocilizumab in Combination With Methotrexate or Other DMARDs: Participants received a weekly SC injection of tocilizumab 162 mg in combination with methotrexate or other non-biologic disease modifying anti-rheumatic drugs (DMARDs) for 52 weeks.
Period: Overall Study
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Started | 22 | 140
Received at Least 1 Dose of Tocilizumab | 21 | 140
Completed | 7 | 65
Not Completed | 15 | 75
Not completed — Other | 11 | 66
Not completed — Protocol Violation | 0 | 1
Not completed — Participant/legal guardian decision | 1 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS population included all participants who received at least one dose of SC tocilizumab.
Groups:
- Tocilizumab Monotherapy: Participants received a weekly SC injection of tocilizumab 162 mg as monotherapy for 52 weeks.
- Tocilizumab in Combination With Methotrexate or Other DMARDs: Participants received a weekly SC injection of tocilizumab 162 mg in combination with methotrexate or other non-biologic DMARDs for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs | Total
Number analyzed (Participants) | 21 | 140 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.63) | 55.3 (10.76) | 55.1 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 104 | 120
  Male | 5 | 36 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 2
Description: DAS28 was calculated from swollen joint count (SJC) and tender joint count (TJC) using 28 joints count, erythrocyte sedimentation rate (ESR; millimeters per hour [mm/hour]), and patient's global assessment of disease activity (measured on a 0 to 100 mm Visual Analog Scale [VAS] where 0 mm=no disease activity and 100 mm=worst disease activity). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. Total score range: 0-10, higher score=higher disease activity. DAS28-ESR greater than or equal to (≥) 2.6 to less than or equal to (≤) 3.2 implied low disease activity, greater than (>) 3.2 to ≤5.1 implied moderate disease activity, >5.1 implied high/severe disease, and less than (<) 2.6 implied clinical remission.
Time Frame: Baseline, Week 2
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 139
units on a scale
  Baseline | 5.52 (1.014) | 5.53 (1.257)
  Change at Week 2: number analyzed (Participants) | 21 | 137
  Change at Week 2 | -1.41 (0.994) | -1.22 (1.131)

2. Primary Outcome: Change From Baseline in DAS28-ESR at Week 4
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and patient's global assessment of disease activity (measured on a 0 to 100 mm VAS where 0 mm=no disease activity and 100 mm=worst disease activity). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. Total score range: 0-10, higher score=higher disease activity. DAS28-ESR ≥2.6 to ≤3.2 implied low disease activity, >3.2 to ≤5.1 implied moderate disease activity, >5.1 implied high/severe disease, and <2.6 implied clinical remission.
Time Frame: Baseline, Week 4
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 137
units on a scale | -1.86 (1.016) | -2.11 (1.215)

3. Primary Outcome: Change From Baseline in DAS28-ESR at Week 8
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 18 | 131
units on a scale | -2.42 (1.352) | -2.62 (1.482)

4. Primary Outcome: Change From Baseline in DAS28-ESR at Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 19 | 128
units on a scale | -2.33 (1.522) | -2.99 (1.510)

5. Primary Outcome: Change From Baseline in DAS28-ESR at Week 16
Description: as for outcome 2
Time Frame: Baseline, Week 16
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 18 | 125
units on a scale | -2.93 (1.218) | -3.07 (1.532)

6. Primary Outcome: Change From Baseline in DAS28-ESR at Week 20
Description: as for outcome 2
Time Frame: Baseline, Week 20
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 19 | 121
units on a scale | -3.17 (1.346) | -3.13 (1.525)

7. Primary Outcome: Change From Baseline in DAS28-ESR at Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 19 | 117
units on a scale | -3.28 (1.379) | -3.33 (1.470)

8. Primary Outcome: Change From Baseline in DAS28-ESR at Week 28
Description: as for outcome 2
Time Frame: Baseline, Week 28
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 19 | 115
units on a scale | -3.54 (1.260) | -3.32 (1.552)

9. Primary Outcome: Change From Baseline in DAS28-ESR at Week 32
Description: as for outcome 2
Time Frame: Baseline, Week 32
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 19 | 115
units on a scale | -3.19 (1.418) | -3.54 (1.448)

10. Primary Outcome: Change From Baseline in DAS28-ESR at Week 36
Description: as for outcome 2
Time Frame: Baseline, Week 36
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 18 | 114
units on a scale | -3.57 (1.358) | -3.55 (1.589)

11. Primary Outcome: Change From Baseline in DAS28-ESR at Week 40
Description: as for outcome 2
Time Frame: Baseline, Week 40
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 17 | 111
units on a scale | -3.82 (1.143) | -3.64 (1.524)

12. Primary Outcome: Change From Baseline in DAS28-ESR at Week 44
Description: as for outcome 2
Time Frame: Baseline, Week 44
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 17 | 107
units on a scale | -3.61 (1.325) | -3.65 (1.574)

13. Primary Outcome: Change From Baseline in DAS28-ESR at Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 16 | 107
units on a scale | -3.54 (1.146) | -3.65 (1.552)

14. Primary Outcome: Change From Baseline in DAS28-ESR at Week 52
Description: as for outcome 2
Time Frame: Baseline, Week 52
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 15 | 107
units on a scale | -3.75 (1.361) | -3.67 (1.592)

15. Primary Outcome: Change From Baseline in DAS28-ESR at Early Withdrawal
Description: as for outcome 2
Time Frame: Baseline, early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 5 | 28
units on a scale | -2.88 (1.236) | -1.63 (1.480)

16. Secondary Outcome: Number of Participants Achieving an American College of Rheumatology Criteria 20 (ACR20) Response
Description: A participant had an ACR20 response if there was at least a 20 percent (%) improvement, ie, reduction from Baseline, in TJC (68 joints) and SJC (66 joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, averaged to 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either C-reactive protein [CRP] or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 6 | 23
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 6 | 68
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 11 | 69
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 10 | 83
  Week 16: number analyzed (Participants) | 19 | 125
  Week 16 | 13 | 83
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 15 | 86
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 15 | 90
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 14 | 87
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 13 | 89
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 12 | 92
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 13 | 91
  Week 44: number analyzed (Participants) | 17 | 108
  Week 44 | 12 | 88
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 12 | 87
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 12 | 88
  Early withdrawal: number analyzed (Participants) | 5 | 29
  Early withdrawal | 3 | 10

17. Secondary Outcome: Number of Participants Achieving an ACR50 Response
Description: A participant had an ACR50 response if there was at least a 50% improvement, ie, reduction from Baseline, in TJC (68 joints) and SJC (66 joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, averaged to 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 0 | 5
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 3 | 20
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 6 | 43
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 8 | 54
  Week 16: number analyzed (Participants) | 19 | 125
  Week 16 | 7 | 62
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 9 | 61
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 9 | 64
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 13 | 68
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 8 | 69
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 9 | 74
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 9 | 71
  Week 44: number analyzed (Participants) | 17 | 108
  Week 44 | 10 | 72
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 11 | 73
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 8 | 73
  Early withdrawal: number analyzed (Participants) | 5 | 29
  Early withdrawal | 2 | 4

18. Secondary Outcome: Number of Participants Achieving an ACR70 Response
Description: A participant had an ACR70 response if there was at least a 70% improvement, ie, reduction from Baseline, in TJC (68 joints) and SJC (66 joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0 mm=no disease activity to 100 mm=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0 mm=no pain to 100 mm=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, averaged to 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 0 | 0
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 1 | 9
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 4 | 19
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 3 | 30
  Week 16: number analyzed (Participants) | 19 | 125
  Week 16 | 3 | 32
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 7 | 37
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 5 | 38
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 6 | 44
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 6 | 47
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 7 | 48
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 8 | 49
  Week 44: number analyzed (Participants) | 17 | 108
  Week 44 | 6 | 53
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 8 | 56
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 7 | 54
  Early withdrawal: number analyzed (Participants) | 5 | 29
  Early withdrawal | 2 | 1

19. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response (Good, Moderate or No Response) Based on DAS28-ESR
Description: DAS28-ESR was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and patient's global assessment of disease activity (VAS: 0 mm=no disease activity to 100 mm=maximum disease activity). DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. The DAS28-ESR based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline >1.2 with a DAS28 score ≤3.2; moderate responders had a change from baseline >1.2 with a DAS28 score >3.2 or a change from baseline >0.6 to ≤1.2 with a DAS28 score ≤5.1. Participants with change from baseline >0.6 to ≤1.2 with a DAS28 score >5.1, or any score with change from baseline ≤0.6, were assessed as non-responders.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Week 2: No response: number analyzed (Participants) | 21 | 137
  Week 2: No response | 4 | 56
  Week 2: Moderate response: number analyzed (Participants) | 21 | 137
  Week 2: Moderate response | 10 | 56
  Week 2: Good response: number analyzed (Participants) | 21 | 137
  Week 2: Good response | 7 | 25
  Week 4: No response: number analyzed (Participants) | 21 | 137
  Week 4: No response | 3 | 22
  Week 4: Moderate response: number analyzed (Participants) | 21 | 137
  Week 4: Moderate response | 7 | 58
  Week 4: Good response: number analyzed (Participants) | 21 | 137
  Week 4: Good response | 11 | 57
  Week 8: No response: number analyzed (Participants) | 18 | 131
  Week 8: No response | 1 | 11
  Week 8: Moderate response: number analyzed (Participants) | 18 | 131
  Week 8: Moderate response | 9 | 48
  Week 8: Good response: number analyzed (Participants) | 18 | 131
  Week 8: Good response | 8 | 72
  Week 12: No response: number analyzed (Participants) | 19 | 128
  Week 12: No response | 4 | 11
  Week 12: Moderate response: number analyzed (Participants) | 19 | 128
  Week 12: Moderate response | 3 | 34
  Week 12: Good response: number analyzed (Participants) | 19 | 128
  Week 12: Good response | 12 | 83
  Week 16: No response: number analyzed (Participants) | 18 | 125
  Week 16: No response | 1 | 9
  Week 16: Moderate response: number analyzed (Participants) | 18 | 125
  Week 16: Moderate response | 4 | 30
  Week 16: Good response: number analyzed (Participants) | 18 | 125
  Week 16: Good response | 13 | 86
  Week 20: No response: number analyzed (Participants) | 19 | 121
  Week 20: No response | 0 | 9
  Week 20: Moderate response: number analyzed (Participants) | 19 | 121
  Week 20: Moderate response | 5 | 27
  Week 20: Good response: number analyzed (Participants) | 19 | 121
  Week 20: Good response | 14 | 85
  Week 24: No response: number analyzed (Participants) | 19 | 117
  Week 24: No response | 1 | 7
  Week 24: Moderate response: number analyzed (Participants) | 19 | 117
  Week 24: Moderate response | 2 | 21
  Week 24: Good response: number analyzed (Participants) | 19 | 117
  Week 24: Good response | 16 | 89
  Week 28: No response: number analyzed (Participants) | 19 | 115
  Week 28: No response | 1 | 5
  Week 28: Moderate response: number analyzed (Participants) | 19 | 115
  Week 28: Moderate response | 0 | 24
  Week 28: Good response: number analyzed (Participants) | 19 | 115
  Week 28: Good response | 18 | 86
  Week 32: No response: number analyzed (Participants) | 19 | 115
  Week 32: No response | 1 | 3
  Week 32: Moderate response: number analyzed (Participants) | 19 | 115
  Week 32: Moderate response | 2 | 21
  Week 32: Good response: number analyzed (Participants) | 19 | 115
  Week 32: Good response | 16 | 91
  Week 36: No response: number analyzed (Participants) | 18 | 114
  Week 36: No response | 0 | 4
  Week 36: Moderate response: number analyzed (Participants) | 18 | 114
  Week 36: Moderate response | 3 | 19
  Week 36: Good response: number analyzed (Participants) | 18 | 114
  Week 36: Good response | 15 | 91
  Week 40: No response: number analyzed (Participants) | 17 | 111
  Week 40: No response | 0 | 2
  Week 40: Moderate response: number analyzed (Participants) | 17 | 111
  Week 40: Moderate response | 1 | 15
  Week 40: Good response: number analyzed (Participants) | 17 | 111
  Week 40: Good response | 16 | 94
  Week 44: No response: number analyzed (Participants) | 17 | 107
  Week 44: No response | 0 | 5
  Week 44: Moderate response: number analyzed (Participants) | 17 | 107
  Week 44: Moderate response | 2 | 15
  Week 44: Good response: number analyzed (Participants) | 17 | 107
  Week 44: Good response | 15 | 87
  Week 48: No response: number analyzed (Participants) | 16 | 107
  Week 48: No response | 0 | 4
  Week 48: Moderate response: number analyzed (Participants) | 16 | 107
  Week 48: Moderate response | 2 | 13
  Week 48: Good response: number analyzed (Participants) | 16 | 107
  Week 48: Good response | 14 | 90
  Week 52: No response: number analyzed (Participants) | 15 | 107
  Week 52: No response | 0 | 5
  Week 52: Moderate response: number analyzed (Participants) | 15 | 107
  Week 52: Moderate response | 3 | 12
  Week 52: Good response: number analyzed (Participants) | 15 | 107
  Week 52: Good response | 12 | 90
  Early Withdrawal: No response: number analyzed (Participants) | 5 | 28
  Early Withdrawal: No response | 0 | 11
  Early Withdrawal: Moderate response: number analyzed (Participants) | 5 | 28
  Early Withdrawal: Moderate response | 1 | 8
  Early Withdrawal: Good response: number analyzed (Participants) | 5 | 28
  Early Withdrawal: Good response | 4 | 9

20. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at Early Withdrawal
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, patient and physician global assessment of disease activity assessed on 0-10 centimeter (cm) VAS (0 cm= no disease activity and 10 cm= worst disease activity), and CRP in milligrams per liter (mg/L). SDAI total score = 0-86. SDAI ≤3.3 indicates clinical remission, >3.3 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 136
units on a scale
  Baseline | 31.23 (11.892) | 32.33 (11.620)
  Change at Week 2: number analyzed (Participants) | 21 | 132
  Change at Week 2 | -9.80 (10.406) | -6.94 (9.710)
  Change at Week 4: number analyzed (Participants) | 19 | 131
  Change at Week 4 | -12.64 (10.502) | -13.92 (10.666)
  Change at Week 8: number analyzed (Participants) | 17 | 127
  Change at Week 8 | -19.75 (12.978) | -17.21 (12.900)
  Change at Week 12: number analyzed (Participants) | 16 | 120
  Change at Week 12 | -14.65 (15.003) | -20.26 (12.739)
  Change at Week 16: number analyzed (Participants) | 16 | 118
  Change at Week 16 | -19.48 (9.649) | -21.16 (11.945)
  Change at Week 20: number analyzed (Participants) | 18 | 115
  Change at Week 20 | -23.67 (14.015) | -20.50 (11.630)
  Change at Week 24: number analyzed (Participants) | 19 | 112
  Change at Week 24 | -24.31 (13.469) | -23.48 (12.417)
  Change at Week 28: number analyzed (Participants) | 19 | 109
  Change at Week 28 | -24.87 (12.554) | -23.26 (12.418)
  Change at Week 32: number analyzed (Participants) | 19 | 109
  Change at Week 32 | -22.98 (12.850) | -24.94 (11.399)
  Change at Week 36: number analyzed (Participants) | 18 | 107
  Change at Week 36 | -26.32 (12.795) | -24.65 (11.268)
  Change at Week 40: number analyzed (Participants) | 17 | 106
  Change at Week 40 | -27.29 (13.280) | -25.46 (12.210)
  Change at Week 44: number analyzed (Participants) | 16 | 101
  Change at Week 44 | -27.71 (12.851) | -26.08 (11.835)
  Change at Week 48: number analyzed (Participants) | 16 | 102
  Change at Week 48 | -26.83 (13.615) | -26.13 (11.189)
  Change at Week 52: number analyzed (Participants) | 15 | 104
  Change at Week 52 | -27.45 (14.351) | -26.15 (12.791)
  Change at early withdrawal: number analyzed (Participants) | 5 | 28
  Change at early withdrawal | -18.94 (14.681) | -9.45 (12.533)

21. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at Early Withdrawal
Description: The CDAI is the numerical sum of four outcome parameters: TJC and SJC based on a 28-joint assessment, patient and physician's global assessment of disease activity assessed on 0-10 cm VAS (0 cm= no disease activity and 10 cm= worst disease activity). CDAI total score = 0-76. CDAI ≤2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 139
units on a scale
  Baseline | 29.69 (11.209) | 30.88 (10.953)
  Change at Week 2: number analyzed (Participants) | 21 | 137
  Change at Week 2 | -8.35 (10.433) | -5.16 (9.323)
  Change at Week 4: number analyzed (Participants) | 21 | 137
  Change at Week 4 | -11.87 (10.062) | -12.26 (10.137)
  Change at Week 8: number analyzed (Participants) | 18 | 130
  Change at Week 8 | -17.74 (12.289) | -15.63 (11.873)
  Change at Week 12: number analyzed (Participants) | 19 | 128
  Change at Week 12 | -15.39 (14.216) | -18.66 (11.895)
  Change at Week 16: number analyzed (Participants) | 19 | 125
  Change at Week 16 | -20.70 (11.694) | -19.51 (11.124)
  Change at Week 20: number analyzed (Participants) | 18 | 121
  Change at Week 20 | -22.19 (13.545) | -19.23 (11.433)
  Change at Week 24: number analyzed (Participants) | 19 | 117
  Change at Week 24 | -22.88 (12.720) | -21.96 (11.825)
  Change at Week 28: number analyzed (Participants) | 19 | 115
  Change at Week 28 | -23.43 (11.573) | -21.48 (11.585)
  Change at Week 32: number analyzed (Participants) | 19 | 115
  Change at Week 32 | -21.55 (12.019) | -23.20 (10.842)
  Change at Week 36: number analyzed (Participants) | 18 | 114
  Change at Week 36 | -24.86 (11.854) | -23.10 (11.263)
  Change at Week 40: number analyzed (Participants) | 17 | 111
  Change at Week 40 | -25.74 (12.488) | -24.01 (11.282)
  Change at Week 44: number analyzed (Participants) | 17 | 106
  Change at Week 44 | -25.42 (11.971) | -24.42 (11.186)
  Change at Week 48: number analyzed (Participants) | 16 | 106
  Change at Week 48 | -25.36 (12.718) | -24.59 (10.645)
  Change at Week 52: number analyzed (Participants) | 16 | 107
  Change at Week 52 | -25.48 (13.049) | -24.42 (12.599)
  Change at early withdrawal: number analyzed (Participants) | 5 | 29
  Change at early withdrawal | -17.78 (14.667) | -8.68 (11.909)

22. Secondary Outcome: Percent Change From Baseline in Total TJC on 68 Joints at Week 52
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 68. A reduction in number of tender joints compared to baseline indicates improvement. The outcome is reported as the percent change from baseline to end of treatment (52 weeks).
Time Frame: Baseline, Week 52
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 15 | 106
percent change | -83.12 (26.607) | -80.44 (41.226)

23. Secondary Outcome: Change From Baseline in Total TJC on 28 Joints at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at Early Withdrawal
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28. A reduction in number of tender joints compared to baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 139
tender joints
  Baseline | 10.4 (6.46) | 12.9 (7.06)
  Change at Week 2: number analyzed (Participants) | 21 | 137
  Change at Week 2 | -3.4 (5.62) | -2.4 (5.63)
  Change at Week 4: number analyzed (Participants) | 21 | 137
  Change at Week 4 | -3.9 (5.80) | -5.4 (6.14)
  Change at Week 8: number analyzed (Participants) | 18 | 132
  Change at Week 8 | -6.6 (6.41) | -6.4 (6.94)
  Change at Week 12: number analyzed (Participants) | 19 | 128
  Change at Week 12 | -6.0 (6.71) | -8.0 (7.35)
  Change at Week 16: number analyzed (Participants) | 19 | 125
  Change at Week 16 | -7.9 (6.35) | -8.2 (7.05)
  Change at Week 20: number analyzed (Participants) | 19 | 122
  Change at Week 20 | -8.5 (6.59) | -8.3 (7.09)
  Change at Week 24: number analyzed (Participants) | 19 | 117
  Change at Week 24 | -8.3 (7.41) | -9.3 (7.53)
  Change at Week 28: number analyzed (Participants) | 19 | 115
  Change at Week 28 | -8.7 (6.26) | -9.2 (7.04)
  Change at Week 32: number analyzed (Participants) | 19 | 115
  Change at Week 32 | -7.6 (6.64) | -10.1 (6.76)
  Change at Week 36: number analyzed (Participants) | 18 | 114
  Change at Week 36 | -9.4 (6.25) | -9.7 (7.23)
  Change at Week 40: number analyzed (Participants) | 17 | 111
  Change at Week 40 | -10.1 (6.64) | -10.3 (6.74)
  Change at Week 44: number analyzed (Participants) | 17 | 108
  Change at Week 44 | -9.7 (6.46) | -10.4 (6.63)
  Change at Week 48: number analyzed (Participants) | 16 | 107
  Change at Week 48 | -9.6 (6.36) | -10.5 (6.70)
  Change at Week 52: number analyzed (Participants) | 16 | 107
  Change at Week 52 | -9.4 (7.15) | -10.4 (8.01)
  Change at early withdrawal: number analyzed (Participants) | 5 | 29
  Change at early withdrawal | -7.0 (6.24) | -3.3 (7.46)

24. Secondary Outcome: Percent Change From Baseline in Total SJC on 66 Joints at Week 52
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 66. A reduction in number of swollen joints compared to baseline indicates improvement. The outcome is reported as the percent change from baseline to end of treatment (52 weeks).
Time Frame: Baseline, Week 52
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 16 | 102
percent change | -89.31 (20.059) | -74.77 (66.277)

25. Secondary Outcome: Change From Baseline in Total SJC on 28 Joints at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at Early Withdrawal
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28. A reduction in number of swollen joints compared to baseline indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 139
swollen joints
  Baseline | 7.0 (4.64) | 5.6 (4.43)
  Change at Week 2: number analyzed (Participants) | 21 | 137
  Change at Week 2 | -2.5 (4.31) | -0.8 (3.95)
  Change at Week 4: number analyzed (Participants) | 21 | 137
  Change at Week 4 | -4.2 (3.79) | -2.5 (3.81)
  Change at Week 8: number analyzed (Participants) | 18 | 132
  Change at Week 8 | -4.8 (4.21) | -3.2 (4.40)
  Change at Week 12: number analyzed (Participants) | 19 | 128
  Change at Week 12 | -4.2 (4.37) | -3.8 (4.36)
  Change at Week 16: number analyzed (Participants) | 19 | 125
  Change at Week 16 | -5.3 (4.67) | -3.9 (4.41)
  Change at Week 20: number analyzed (Participants) | 19 | 122
  Change at Week 20 | -5.6 (5.08) | -4.2 (4.60)
  Change at Week 24: number analyzed (Participants) | 19 | 117
  Change at Week 24 | -5.9 (5.12) | -4.7 (4.21)
  Change at Week 28: number analyzed (Participants) | 19 | 115
  Change at Week 28 | -6.4 (4.90) | -4.4 (4.63)
  Change at Week 32: number analyzed (Participants) | 19 | 115
  Change at Week 32 | -5.4 (5.10) | -4.8 (4.37)
  Change at Week 36: number analyzed (Participants) | 18 | 114
  Change at Week 36 | -6.5 (4.57) | -4.9 (4.41)
  Change at Week 40: number analyzed (Participants) | 17 | 111
  Change at Week 40 | -6.6 (5.12) | -5.0 (4.82)
  Change at Week 44: number analyzed (Participants) | 17 | 108
  Change at Week 44 | -6.6 (5.28) | -5.2 (4.71)
  Change at Week 48: number analyzed (Participants) | 16 | 107
  Change at Week 48 | -6.4 (4.83) | -5.0 (4.48)
  Change at Week 52: number analyzed (Participants) | 16 | 107
  Change at Week 52 | -6.3 (4.81) | -5.1 (4.51)
  Change at early withdrawal: number analyzed (Participants) | 5 | 29
  Change at early withdrawal | -5.8 (5.59) | -1.7 (4.43)

26. Secondary Outcome: Number of Participants Who Achieved Low Disease Activity as Defined by DAS28-ESR ≤3.2
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and patient's global assessment of disease activity (measured on a 0 to 100 mm VAS where 0 mm=no disease activity and 100 mm=worst disease activity). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. Total score range: 0-10, higher score=higher disease activity. DAS28-ESR ≥2.6 to ≤3.2 implied low disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 0 | 5
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 7 | 18
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 9 | 30
  Week 8: number analyzed (Participants) | 18 | 131
  Week 8 | 3 | 25
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 6 | 23
  Week 16: number analyzed (Participants) | 18 | 125
  Week 16 | 3 | 20
  Week 20: number analyzed (Participants) | 19 | 121
  Week 20 | 3 | 15
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 2 | 15
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 4 | 15
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 5 | 14
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 1 | 14
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 3 | 14
  Week 44: number analyzed (Participants) | 17 | 107
  Week 44 | 5 | 10
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 3 | 12
  Week 52: number analyzed (Participants) | 15 | 107
  Week 52 | 0 | 11
  Early withdrawal: number analyzed (Participants) | 5 | 29
  Early withdrawal | 2 | 4

27. Secondary Outcome: Number of Participants Who Achieved Remission as Defined by DAS28-ESR <2.6
Description: DAS28 was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and patient's global assessment of disease activity (measured on a 0 to 100 mm VAS where 0 mm=no disease activity and 100 mm=worst disease activity). DAS28 scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. Total score range: 0-10, higher score=higher disease activity. DAS28-ESR <2.6 implied clinical remission.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 0 | 3
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 1 | 15
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 2 | 34
  Week 8: number analyzed (Participants) | 18 | 131
  Week 8 | 5 | 53
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 6 | 66
  Week 16: number analyzed (Participants) | 18 | 125
  Week 16 | 10 | 72
  Week 20: number analyzed (Participants) | 19 | 121
  Week 20 | 11 | 75
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 14 | 76
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 14 | 73
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 12 | 80
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 14 | 80
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 13 | 81
  Week 44: number analyzed (Participants) | 17 | 107
  Week 44 | 10 | 80
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 11 | 78
  Week 52: number analyzed (Participants) | 15 | 107
  Week 52 | 12 | 80
  Early withdrawal: number analyzed (Participants) | 5 | 29
  Early withdrawal | 3 | 7

28. Secondary Outcome: Number of Participants With Non-Biologic DMARD/Corticosteroid Dose Reductions and/or Discontinuation
Description: Results are reported for number of participants who had non-biologic DMARD/corticosteroid dose reductions and/or discontinuation by reasons for dose reductions or discontinuation (safety reasons, discomfort, lack of efficacy, other reasons, and unknown reasons). Participants may be included under more than one reason.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, at early withdrawal (up to Week 52), follow-up Week 4 (up to Week 56), and follow-up Week 8 (up to Week 60)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Baseline: Safety | 0 | 1
  Baseline: Discomfort | 0 | 0
  Baseline: Lack of efficacy | 0 | 1
  Baseline: Other | 0 | 2
  Baseline: Unknown | 0 | 0
  Week 2: Safety: number analyzed (Participants) | 21 | 137
  Week 2: Safety | 0 | 4
  Week 2: Discomfort: number analyzed (Participants) | 21 | 137
  Week 2: Discomfort | 0 | 0
  Week 2: Lack of efficacy: number analyzed (Participants) | 21 | 137
  Week 2: Lack of efficacy | 0 | 0
  Week 2: Other: number analyzed (Participants) | 21 | 137
  Week 2: Other | 0 | 7
  Week 2: Unknown: number analyzed (Participants) | 21 | 137
  Week 2: Unknown | 0 | 0
  Week 4: Safety: number analyzed (Participants) | 21 | 137
  Week 4: Safety | 0 | 6
  Week 4: Discomfort: number analyzed (Participants) | 21 | 137
  Week 4: Discomfort | 0 | 0
  Week 4: Lack of efficacy: number analyzed (Participants) | 21 | 137
  Week 4: Lack of efficacy | 0 | 1
  Week 4: Other: number analyzed (Participants) | 21 | 137
  Week 4: Other | 1 | 9
  Week 4: Unknown: number analyzed (Participants) | 21 | 137
  Week 4: Unknown | 0 | 1
  Week 8: Safety: number analyzed (Participants) | 18 | 132
  Week 8: Safety | 0 | 8
  Week 8: Discomfort: number analyzed (Participants) | 18 | 132
  Week 8: Discomfort | 0 | 0
  Week 8: Lack of efficacy: number analyzed (Participants) | 18 | 132
  Week 8: Lack of efficacy | 0 | 0
  Week 8: Other: number analyzed (Participants) | 18 | 132
  Week 8: Other | 1 | 13
  Week 8: Unknown: number analyzed (Participants) | 18 | 132
  Week 8: Unknown | 0 | 1
  Week 12: Safety: number analyzed (Participants) | 19 | 128
  Week 12: Safety | 0 | 6
  Week 12: Discomfort 8: number analyzed (Participants) | 19 | 128
  Week 12: Discomfort 8 | 0 | 2
  Week 12: Lack of efficacy: number analyzed (Participants) | 19 | 128
  Week 12: Lack of efficacy | 0 | 0
  Week 12: Other: number analyzed (Participants) | 19 | 128
  Week 12: Other | 2 | 14
  Week 12: Unknown: number analyzed (Participants) | 19 | 128
  Week 12: Unknown | 0 | 0
  Week 16: Safety: number analyzed (Participants) | 19 | 126
  Week 16: Safety | 0 | 7
  Week 16: Discomfort: number analyzed (Participants) | 19 | 126
  Week 16: Discomfort | 0 | 0
  Week 16: Lack of efficacy: number analyzed (Participants) | 19 | 126
  Week 16: Lack of efficacy | 0 | 1
  Week 16: Other: number analyzed (Participants) | 19 | 126
  Week 16: Other | 2 | 13
  Week 16: Unknown: number analyzed (Participants) | 19 | 126
  Week 16: Unknown | 0 | 0
  Week 20: Safety: number analyzed (Participants) | 19 | 122
  Week 20: Safety | 0 | 6
  Week 20: Discomfort: number analyzed (Participants) | 19 | 122
  Week 20: Discomfort | 0 | 0
  Week 20: Lack of efficacy: number analyzed (Participants) | 19 | 122
  Week 20: Lack of efficacy | 0 | 0
  Week 20: Other: number analyzed (Participants) | 19 | 122
  Week 20: Other | 2 | 9
  Week 20: Unknown: number analyzed (Participants) | 19 | 122
  Week 20: Unknown | 0 | 1
  Week 24: Safety: number analyzed (Participants) | 19 | 117
  Week 24: Safety | 0 | 5
  Week 24:Discomfort: number analyzed (Participants) | 19 | 117
  Week 24:Discomfort | 0 | 0
  Week 24: Lack of efficacy: number analyzed (Participants) | 19 | 117
  Week 24: Lack of efficacy | 0 | 0
  Week 24: Other: number analyzed (Participants) | 19 | 117
  Week 24: Other | 1 | 13
  Week 24: Unknown: number analyzed (Participants) | 19 | 117
  Week 24: Unknown | 0 | 1
  Week 28: Safety: number analyzed (Participants) | 19 | 116
  Week 28: Safety | 0 | 3
  Week 28: Discomfort: number analyzed (Participants) | 19 | 116
  Week 28: Discomfort | 0 | 0
  Week 28: Lack of efficacy: number analyzed (Participants) | 19 | 116
  Week 28: Lack of efficacy | 0 | 1
  Week 28: Other: number analyzed (Participants) | 19 | 116
  Week 28: Other | 1 | 7
  Week 28: Unknown: number analyzed (Participants) | 19 | 116
  Week 28: Unknown | 0 | 0
  Week 32: Safety: number analyzed (Participants) | 19 | 115
  Week 32: Safety | 0 | 4
  Week 32: Discomfort: number analyzed (Participants) | 19 | 115
  Week 32: Discomfort | 0 | 0
  Week 32: Lack of efficacy: number analyzed (Participants) | 19 | 115
  Week 32: Lack of efficacy | 0 | 2
  Week 32: Other: number analyzed (Participants) | 19 | 115
  Week 32: Other | 1 | 11
  Week 32: Unknown: number analyzed (Participants) | 19 | 115
  Week 32: Unknown | 0 | 0
  Week 36: Safety: number analyzed (Participants) | 18 | 114
  Week 36: Safety | 0 | 3
  Week 36: Discomfort: number analyzed (Participants) | 18 | 114
  Week 36: Discomfort | 0 | 1
  Week 36: Lack of efficacy: number analyzed (Participants) | 18 | 114
  Week 36: Lack of efficacy | 0 | 0
  Week 36: Other: number analyzed (Participants) | 18 | 114
  Week 36: Other | 2 | 3
  Week 36: Unknown: number analyzed (Participants) | 18 | 114
  Week 36: Unknown | 0 | 0
  Week 40: Safety: number analyzed (Participants) | 17 | 111
  Week 40: Safety | 0 | 4
  Week 40: Discomfort: number analyzed (Participants) | 17 | 111
  Week 40: Discomfort | 0 | 1
  Week 40: Lack of efficacy: number analyzed (Participants) | 17 | 111
  Week 40: Lack of efficacy | 0 | 1
  Week 40: Other: number analyzed (Participants) | 17 | 111
  Week 40: Other | 1 | 1
  Week 40: Unknown: number analyzed (Participants) | 17 | 111
  Week 40: Unknown | 0 | 0
  Week 44: Safety: number analyzed (Participants) | 17 | 108
  Week 44: Safety | 0 | 3
  Week 44: Discomfort: number analyzed (Participants) | 17 | 108
  Week 44: Discomfort | 0 | 0
  Week 44: Lack of efficacy: number analyzed (Participants) | 17 | 108
  Week 44: Lack of efficacy | 0 | 0
  Week 44: Other: number analyzed (Participants) | 17 | 108
  Week 44: Other | 0 | 7
  Week 44: Unknown: number analyzed (Participants) | 17 | 108
  Week 44: Unknown | 0 | 0
  Week 48: Safety: number analyzed (Participants) | 16 | 107
  Week 48: Safety | 0 | 3
  Week 48: Discomfort: number analyzed (Participants) | 16 | 107
  Week 48: Discomfort | 0 | 0
  Week 48: Lack of efficacy: number analyzed (Participants) | 16 | 107
  Week 48: Lack of efficacy | 0 | 1
  Week 48: Other: number analyzed (Participants) | 16 | 107
  Week 48: Other | 1 | 3
  Week 48: Unknown: number analyzed (Participants) | 16 | 107
  Week 48: Unknown | 0 | 0
  Week 52: Safety: number analyzed (Participants) | 16 | 107
  Week 52: Safety | 0 | 0
  Week 52: Discomfort: number analyzed (Participants) | 16 | 107
  Week 52: Discomfort | 0 | 0
  Week 52: Lack of efficacy: number analyzed (Participants) | 16 | 107
  Week 52: Lack of efficacy | 0 | 0
  Week 52: Other: number analyzed (Participants) | 16 | 107
  Week 52: Other | 0 | 1
  Week 52: Unknown: number analyzed (Participants) | 16 | 107
  Week 52: Unknown | 0 | 0
  Early withdrawal: Safety: number analyzed (Participants) | 5 | 30
  Early withdrawal: Safety | 0 | 0
  Early withdrawal: Discomfort: number analyzed (Participants) | 5 | 30
  Early withdrawal: Discomfort | 0 | 0
  Early withdrawal: Lack of efficacy: number analyzed (Participants) | 5 | 30
  Early withdrawal: Lack of efficacy | 0 | 0
  Early withdrawal: Other: number analyzed (Participants) | 5 | 30
  Early withdrawal: Other | 1 | 8
  Early withdrawal: Unknown: number analyzed (Participants) | 5 | 30
  Early withdrawal: Unknown | 0 | 0
  Follow-up Week 4: Safety: number analyzed (Participants) | 8 | 70
  Follow-up Week 4: Safety | 0 | 0
  Follow-up Week 4: Discomfort: number analyzed (Participants) | 8 | 70
  Follow-up Week 4: Discomfort | 0 | 0
  Follow-up Week 4: Lack of efficacy: number analyzed (Participants) | 8 | 70
  Follow-up Week 4: Lack of efficacy | 0 | 0
  Follow-up Week 4: Other: number analyzed (Participants) | 8 | 70
  Follow-up Week 4: Other | 0 | 2
  Follow-up Week 4: Unknown: number analyzed (Participants) | 8 | 70
  Follow-up Week 4: Unknown | 0 | 1
  Follow-up Week 8: Safety: number analyzed (Participants) | 9 | 65
  Follow-up Week 8: Safety | 0 | 0
  Follow-up Week 8: Discomfort: number analyzed (Participants) | 9 | 65
  Follow-up Week 8: Discomfort | 0 | 0
  Follow-up Week 8: Lack of efficacy: number analyzed (Participants) | 9 | 65
  Follow-up Week 8: Lack of efficacy | 0 | 0
  Follow-up Week 8: Other: number analyzed (Participants) | 9 | 65
  Follow-up Week 8: Other | 0 | 0
  Follow-up Week 8: Unknown: number analyzed (Participants) | 9 | 65
  Follow-up Week 8: Unknown | 0 | 0

29. Secondary Outcome: Percentage of Methotrexate Adherence as Assessed by Methotrexate Adherence Questionnaire
Description: Methotrexate adherence was determined from responses to the question 'Over the last 3 months you were prescribed 12 doses of methotrexate, how many (approximately) have you taken?' Adherence (%) was calculated as: (Approximate number of doses taken/12)*100.
Time Frame: Baseline, Weeks 12, 24, 36, 52, and at early withdrawal (up to Week 52)
Population: FAS population. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome. Results are provided for single arm as participants in "Tocilizumab Monotherapy" arm did not receive methotrexate.
Measure: Mean (Standard Deviation); unit: percentage of methotrexate adherence
Arm/Group | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 97
percentage of methotrexate adherence
  Baseline | 96.82 (7.747)
  Week 12: number analyzed (Participants) | 80
  Week 12 | 92.92 (14.412)
  Week 24: number analyzed (Participants) | 65
  Week 24 | 91.54 (20.915)
  Week 36: number analyzed (Participants) | 60
  Week 36 | 90.14 (21.456)
  Week 52: number analyzed (Participants) | 60
  Week 52 | 95.28 (11.417)
  Early withdrawal: number analyzed (Participants) | 17
  Early withdrawal | 90.69 (18.367)

30. Secondary Outcome: Patient Global Assessment of Disease Activity VAS Score
Description: Patient global assessment of disease activity was measured on a 0 to 100 mm horizontal VAS where 0 mm=no disease activity and 100 mm=maximum disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
mm
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 59.6 (26.94) | 62.3 (20.72)
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 50.3 (24.01) | 54.5 (22.12)
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 46.4 (26.43) | 42.3 (23.22)
  Week 8: number analyzed (Participants) | 18 | 131
  Week 8 | 35.8 (24.73) | 36.2 (24.43)
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 41.3 (27.67) | 32.1 (23.91)
  Week 16: number analyzed (Participants) | 19 | 126
  Week 16 | 29.6 (21.59) | 29.2 (22.55)
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 25.7 (23.77) | 29.9 (22.99)
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 23.8 (19.55) | 26.6 (21.92)
  Week 28: number analyzed (Participants) | 19 | 116
  Week 28 | 23.2 (16.47) | 26.7 (23.12)
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 24.0 (17.81) | 24.3 (21.66)
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 24.1 (19.13) | 22.3 (21.86)
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 22.5 (19.31) | 21.4 (20.81)
  Week 44: number analyzed (Participants) | 17 | 107
  Week 44 | 22.7 (20.62) | 22.0 (22.83)
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 22.9 (23.31) | 18.9 (20.57)
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 20.6 (18.96) | 21.4 (23.07)
  Early withdrawal: number analyzed (Participants) | 5 | 30
  Early withdrawal | 30.8 (28.78) | 52.4 (24.88)

31. Secondary Outcome: Patient Pain VAS Score
Description: This assessment represents the participant's assessment of his/her current level of pain on a 100 mm horizontal VAS where 0 mm= no pain to 100 mm= unbearable pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS populations.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
mm
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 50.5 (23.78) | 57.5 (21.06)
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 46.1 (22.43) | 51.1 (22.58)
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 47.0 (26.69) | 42.4 (23.80)
  Week 8: number analyzed (Participants) | 18 | 131
  Week 8 | 37.8 (25.75) | 35.3 (24.30)
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 40.9 (29.56) | 30.8 (23.29)
  Week 16: number analyzed (Participants) | 19 | 126
  Week 16 | 29.7 (20.83) | 26.8 (22.61)
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 27.6 (25.48) | 28.6 (23.74)
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 29.9 (22.76) | 25.2 (22.16)
  Week 28: number analyzed (Participants) | 19 | 116
  Week 28 | 24.8 (19.15) | 25.6 (23.18)
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 25.1 (17.92) | 22.6 (21.30)
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 29.6 (20.03) | 22.1 (21.68)
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 27.6 (22.70) | 20.9 (21.24)
  Week 44: number analyzed (Participants) | 17 | 107
  Week 44 | 26.7 (24.25) | 20.0 (21.26)
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 28.6 (28.98) | 17.6 (19.66)
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 22.4 (19.70) | 19.0 (19.83)
  Early withdrawal: number analyzed (Participants) | 5 | 30
  Early withdrawal | 30.4 (29.57) | 51.6 (26.03)

32. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire measures functional status (disability) and health-related quality of life. It measures the participant's ability to perform everyday tasks. The index consists of 20 questions regarding the function of the upper and lower extremities. These questions are summarized in 8 categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common activities over past week. Each question is evaluated according to the degree of severity on a 4-point scale. Total score for HAQ-DI was the average of all questions and ranges from 0 = without any difficulty to 3 = unable to do.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
units on a scale
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 1.806 (0.5551) | 1.738 (0.6406)
  Week 2: number analyzed (Participants) | 20 | 137
  Week 2 | 1.558 (0.7319) | 1.659 (0.6210)
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 1.616 (0.7720) | 1.546 (0.7351)
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 1.508 (0.7597) | 1.404 (0.8115)
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 1.488 (0.9304) | 1.333 (0.8272)
  Week 16: number analyzed (Participants) | 19 | 126
  Week 16 | 1.351 (0.9586) | 1.312 (0.8621)
  Week 20: number analyzed (Participants) | 19 | 119
  Week 20 | 1.409 (0.9071) | 1.318 (0.8608)
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 1.330 (0.8379) | 1.261 (0.8915)
  Week 28: number analyzed (Participants) | 19 | 116
  Week 28 | 1.330 (0.9412) | 1.221 (0.8730)
  Week 32: number analyzed (Participants) | 19 | 114
  Week 32 | 1.351 (0.8816) | 1.232 (0.8870)
  Week 36: number analyzed (Participants) | 18 | 113
  Week 36 | 1.432 (0.9048) | 1.170 (0.8757)
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 1.479 (0.8975) | 1.199 (0.8908)
  Week 44: number analyzed (Participants) | 17 | 108
  Week 44 | 1.442 (0.9392) | 1.130 (0.9206)
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 1.361 (0.9685) | 1.114 (0.8815)
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 1.338 (0.9796) | 1.154 (0.9187)
  Early withdrawal: number analyzed (Participants) | 5 | 30
  Early withdrawal | 1.252 (1.1232) | 1.756 (0.7820)

33. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: The FACIT-F score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (better score).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
units on a scale
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 18.4 (11.14) | 24.3 (11.55)
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 23.1 (12.37) | 27.9 (11.03)
  Week 4: number analyzed (Participants) | 21 | 136
  Week 4 | 25.1 (12.28) | 30.7 (12.10)
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 30.2 (11.58) | 32.8 (11.91)
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 28.4 (11.71) | 33.7 (11.85)
  Week 16: number analyzed (Participants) | 19 | 126
  Week 16 | 31.3 (13.80) | 34.0 (12.53)
  Week 20: number analyzed (Participants) | 19 | 121
  Week 20 | 33.2 (13.57) | 34.1 (12.05)
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 33.8 (15.28) | 35.3 (10.98)
  Week 28: number analyzed (Participants) | 19 | 115
  Week 28 | 32.9 (12.06) | 35.5 (11.59)
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 34.1 (12.68) | 36.2 (11.32)
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 30.3 (13.62) | 36.8 (11.48)
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 31.7 (12.87) | 37.1 (11.69)
  Week 44: number analyzed (Participants) | 17 | 106
  Week 44 | 31.0 (14.02) | 37.2 (11.75)
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 31.6 (14.63) | 37.9 (11.73)
  Week 52: number analyzed (Participants) | 16 | 106
  Week 52 | 33.4 (14.17) | 38.1 (11.16)
  Early withdrawal: number analyzed (Participants) | 4 | 30
  Early withdrawal | 31.3 (2.63) | 24.5 (12.08)

34. Secondary Outcome: Number of Participants Compliant to Tocilizumab Treatment as Measured by Diary Cards and Return Records
Description: A diary card was provided to participants to record home injections. Participants were asked to return all empty drug supply boxes, unused pre-filled syringe, and diary cards to the clinic at each visit as a measure of drug accountability and participant compliance. A participant was considered compliant if the participant correctly administered all scheduled doses of SC tocilizumab during the assessment period.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at early withdrawal (up to Week 52)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Baseline: number analyzed (Participants) | 21 | 139
  Baseline | 21 | 137
  Week 2: number analyzed (Participants) | 21 | 137
  Week 2 | 20 | 126
  Week 4: number analyzed (Participants) | 21 | 137
  Week 4 | 20 | 132
  Week 8: number analyzed (Participants) | 18 | 132
  Week 8 | 18 | 124
  Week 12: number analyzed (Participants) | 19 | 128
  Week 12 | 18 | 121
  Week 16: number analyzed (Participants) | 19 | 126
  Week 16 | 19 | 120
  Week 20: number analyzed (Participants) | 19 | 122
  Week 20 | 18 | 114
  Week 24: number analyzed (Participants) | 19 | 117
  Week 24 | 16 | 107
  Week 28: number analyzed (Participants) | 19 | 116
  Week 28 | 19 | 112
  Week 32: number analyzed (Participants) | 19 | 115
  Week 32 | 17 | 111
  Week 36: number analyzed (Participants) | 18 | 114
  Week 36 | 17 | 105
  Week 40: number analyzed (Participants) | 17 | 111
  Week 40 | 16 | 104
  Week 44: number analyzed (Participants) | 17 | 108
  Week 44 | 16 | 102
  Week 48: number analyzed (Participants) | 16 | 107
  Week 48 | 13 | 107
  Week 52: number analyzed (Participants) | 16 | 107
  Week 52 | 16 | 98
  Early withdrawal: number analyzed (Participants) | 5 | 30
  Early withdrawal | 4 | 27

35. Secondary Outcome: Number of Participants With Anti-Tocilizumab Antibodies
Time Frame: Baseline, Weeks 12 and 24, at early withdrawal (up to Week 52), and follow-up visit (8 weeks after last dose of tocilizumab, up to 60 weeks)
Population: FAS population.
Measure: Number; unit: participants
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
participants
  Baseline: number analyzed (Participants) | 20 | 138
  Baseline | 3 | 6
  Week 12: number analyzed (Participants) | 1 | 0
  Week 12 | 0 |
  Week 24: number analyzed (Participants) | 19 | 116
  Week 24 | 0 | 2
  Early withdrawal: number analyzed (Participants) | 5 | 27
  Early withdrawal | 0 | 0
  Follow-up visit: number analyzed (Participants) | 3 | 21
  Follow-up visit | 0 | 0

36. Secondary Outcome: Serum Levels of Tocilizumab
Time Frame: as for outcome 35
Population: FAS population.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
micrograms per milliliter (mcg/mL)
  Baseline: number analyzed (Participants) | 20 | 138
  Baseline | 0.0000 (0.0000) | 0.0082 (0.09619)
  Week 12: number analyzed (Participants) | 18 | 125
  Week 12 | 35.3953 (22.69069) | 40.2529 (21.05801)
  Week 24: number analyzed (Participants) | 19 | 115
  Week 24 | 53.0416 (39.06367) | 43.9047 (30.41603)
  Early withdrawal: number analyzed (Participants) | 5 | 25
  Early withdrawal | 44.7160 (38.81521) | 17.6160 (22.92477)
  Follow-up visit: number analyzed (Participants) | 3 | 22
  Follow-up visit | 0.0597 (0.10335) | 2.3123 (7.40931)

37. Secondary Outcome: Serum Levels of Soluble Interleukin-6 Receptors (sIL-6Rs)
Time Frame: as for outcome 35
Population: FAS population.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Number analyzed (Participants) | 21 | 140
nanograms per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 8 | 48
  Baseline | 43.63 (10.947) | 42.40 (12.087)
  Week 12: number analyzed (Participants) | 12 | 57
  Week 12 | 577.42 (175.649) | 548.70 (131.079)
  Week 24: number analyzed (Participants) | 12 | 80
  Week 24 | 602.25 (158.541) | 521.07 (160.464)
  Early withdrawal: number analyzed (Participants) | 4 | 18
  Early withdrawal | 639.75 (99.644) | 327.95 (229.481)
  Follow-up visit: number analyzed (Participants) | 3 | 20
  Follow-up visit | 132.23 (93.048) | 125.07 (211.038)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 60
Description: FAS population
Arm/Group | Tocilizumab Monotherapy | Tocilizumab in Combination With Methotrexate or Other DMARDs
Serious Adverse Events (participants affected / at risk) | 3/21 | 7/140
Other Adverse Events (participants affected / at risk) | 19/21 | 135/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=21) | Tocilizumab in Combination With Methotrexate or Other DMARDs (N=140)
Arthritis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Monotherapy (N=21) | Tocilizumab in Combination With Methotrexate or Other DMARDs (N=140)
Nasopharyngitis (Infections and infestations) | 5 | 33
Lower respiratory tract infection (Infections and infestations) | 6 | 25
Upper respiratory tract infection (Infections and infestations) | 2 | 20
Urinary tract infection (Infections and infestations) | 5 | 16
Oral herpes (Infections and infestations) | 1 | 10
Lower respiratory tract infection viral (Infections and infestations) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 32
Nausea (Gastrointestinal disorders) | 0 | 21
Mouth ulceration (Gastrointestinal disorders) | 1 | 18
Vomiting (Gastrointestinal disorders) | 2 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Alanine aminotransferase increased (Investigations) | 2 | 31
Neutrophil count decreased (Investigations) | 0 | 13
Blood cholesterol increased (Investigations) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 11
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 11
Injection site bruising (General disorders) | 3 | 12
Fatigue (General disorders) | 1 | 12
Injection site erythema (General disorders) | 1 | 11
Influenza like illness (General disorders) | 1 | 8
Peripheral swelling (General disorders) | 1 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 21
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 18
Contusion (Injury, poisoning and procedural complications) | 2 | 13
Fall (Injury, poisoning and procedural complications) | 1 | 14
Laceration (Injury, poisoning and procedural complications) | 0 | 7
Headache (Nervous system disorders) | 4 | 13
Dizziness (Nervous system disorders) | 2 | 8
Migraine (Nervous system disorders) | 1 | 7
Paraesthesia (Nervous system disorders) | 2 | 6
Lethargy (Nervous system disorders) | 0 | 7
Neutropenia (Blood and lymphatic system disorders) | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.